CLINICAL TRIAL: NCT04760158
Title: New Technique For Taping on Patellofemoral Pain Syndrome
Brief Title: Comparison of New Technique Taping and Placebo Taping on Patellofemoral Pain Syndrome: A Randomised Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Phd, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/06/02
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Patello Femoral Syndrome
Keywords: Patella Femoral Pain Syndrome; Exercise; Elastic taping; Pain; Kinesiotaping
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Taping group (Experimental): A new star taping technique and exercises were applied to participants.
  Interventions: Other: Exercise
- Sham Taping Group (Sham Comparator): Sham patellar taping and exercises were applied to participants.
  Interventions: Other: Exercise
- control group (Other): Only exercises were applied to participants.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants of this study exercised strengthening and stretching 3 days a week for 6 weeks

SUMMARY:
We included in this study 42 individuals with patellofemoral pain syndrome. 39 of them were completed six weeks of exercise and other groups. We randomized them into three groups. One group is the star technique which is a new patellar taping technique. Another group is placebo taping and the third group is only the exercise group. Both groups performed exercises three times a week for six weeks. Three groups were assessed with knee and hip muscles strength, shortness, performance tests, pain severity in the activity, night, rest, and knee-buckling, and Kujala Scale before and after 4-week exercises.

DETAILED DESCRIPTION:
Based on previous studies those participants who met the following inclusion criteria were invited to participate in the study: i) insidious onset of anterior knee pain with a duration greater than 4 weeks; ii) pain provoked by at least two of the following situations: prolonged sitting or kneeling, squatting, running, hopping or ascending or descending stairs; iii) age ranged between 18-60 years.

Participants were excluded in cases of the clinical history of patellofemoral dislocation or subluxation; knee osteoarthritis; injury or pain from the hip, lumbar spine, or other knee structures (meniscus, ligaments, bursa, synovial plica, infrapatellar fat); traumatic lesions of soft tissues or previous orthopedic surgery in lower limbs; having received knee injections of corticosteroids or hyaluronic acid; cognition or impaired communication; being involved in an ongoing medical-legal dispute; using Canadien or walker; can not walk independently and having an allergy to taping.

ELIGIBILITY:
Inclusion Criteria:

* insidious onset of anterior knee pain with a duration greater than 4 weeks;
* self-reported patellofemoral pain intensity ≥30 mm on the 100 mm Visual Analogue Scale (VAS)
* pain provoked by at least two of the following situations: prolonged sitting or kneeling, squatting, running, hopping, or ascending or descending stairs;
* age ranged between 18-60 years.

Exclusion Criteria:

* the clinical history of patellofemoral dislocation or subluxation; knee osteoarthritis; injury or pain from the hip, lumbar spine, or other knee structures (meniscus, ligaments, bursa, synovial plica, infrapatellar fat)

  -); traumatic lesions of soft tissues or previous orthopedic surgery in lower limbs; having received knee injections of corticosteroids or hyaluronic acid
* cognition or impaired communication
* being involved in an ongoing medical-legal dispute
* using Canadien or walker; can not walk independently
* having an allergy to taping

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
comparision of the effects of new patellar taping technique and placebo taping on performance | 6 weeks
  we analyzed and compared the performance test outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Tezel Y Şahan, Principal Investigator — Kırıkkale University
Locations (1):
- Kırıkkale University, Kırıkkale, Yahşihan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Effects of exercise combined with whole body vibration in patients with patellofemoral pain syndrome: a randomised-controlled clinical trial. BMC Musculoskelet Disord 21, 582 (2020). — http://bmcmusculoskeletdisord.biomedcentral.com/articles/10.1186/s12891-020-03599-2#citeas
- See also: Systematic Review of the Effect of Taping Techniques on Patellofemoral Pain Syndrome — http://pubmed.ncbi.nlm.nih.gov/28617653/
- See also: The Effect of Kinesio Taping on Anterior Knee Pain Consistent With Patellofemoral Pain Syndrome: A Critically Appraised Topic — http://pubmed.ncbi.nlm.nih.gov/25946512/
- See also: Effects of Posterior X Taping on Movement Quality and Knee Pain Intensity during Forward-Step-Down in Patients with Patellofemoral Pain Syndrome — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC7039014/